CLINICAL TRIAL: NCT01187966
Title: A Phase III, Double-blind, Placebo-controlled Study to Determine the Efficacy and Safety of a Low (50 mg/Day) and High (100 mg/Day) Dose of Safinamide, as add-on Therapy, in Patients With Idiopathic Parkinson's Disease With Motor Fluctuations, Treated With a Stable Dose of Levodopa and Who May be Receiving Concomitant Treatment With Stable Doses of a Dopamine Agonist, and/or an Anticholinergic
Brief Title: Efficacy and Safety of Safinamide (50 and 100mg/Day) Versus Placebo, in Patients With Mid-late Stage Parkinson's Disease
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: Newron Pharmaceuticals SPA (Industry)
Responsible Party: Dr Ravi Anand CMO, Newron Pharmaceuticals
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: NW-1015/016/III/2006
Record Dates: First submitted 2010-05-31; First posted 2010-08-24 (Estimated); Last update posted 2010-08-24 (Estimated); Status verified 2010-08

CONDITIONS: Parkinson's Disease
Keywords: Parkinson's Disease; PD; Levodopa; Patients with idiopathic Parkinson's disease with motor fluctuations
MeSH Terms: conditions — Parkinson Disease | interventions — safinamide

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes

ARMS (3):
- Placebo (Placebo Comparator): Drug: Placebo
  Interventions: Drug: Placebo
- High Dose (100mg/day) (Experimental)
  Interventions: Drug: Safinamide
- Low dose (50mg/day) (Experimental)
  Interventions: Drug: Safinamide

INTERVENTIONS:
Drug: Safinamide
  Arms: Low dose (50mg/day)
Drug: Safinamide
  Arms: High Dose (100mg/day)
Drug: Placebo
  Arms: Placebo

SUMMARY:
The purpose of this study is to evaluate the efficacy and safety of two doses of safinamide (50 and 100 mg/day, p.o.), compared to placebo, as add-on therapy in patients with idiopathic Parkinson's disease with motor fluctuations who are currently receiving a stable dose of levodopa.

ELIGIBILITY:
Inclusion Criteria:

* Patients are male or female, age 30-80 years, inclusive. If female, they must be either post-menopausal for at least 12 months, surgically sterilized or have undergone hysterectomy. Patients older than 80 years, who meet all other entry criteria, will be considered for enrollment, with approval of the Newron Medical Expert.
* Patients must have a diagnosis of idiopathic Parkinson's disease of more than 5 years duration; the diagnosis should be based on medical history and neurological examination. Patients with a duration of Parkinson's disease of at least 3 years, who meet all other entry criteria, will be considered for enrollment, with approval of the CRO Medical Monitor.
* Patients must have a Hoehn and Yahr stage of I-IV during an "off" phase.
* Patients should be levodopa responsive and must have been receiving treatment with a stable dose of levodopa [4-10 doses per day of any levodopa preparation (including CR, IR or a combination of CR/IR), plus benserazide/carbidopa; with or without addition of a COMT inhibitor] and may be receiving concomitant treatment with stable doses of a dopamine agonist and/or an anticholinergic at the screening visit. Patients will receive the study medication as add-on therapy starting at baseline.
* Patients should have motor fluctuations, with >1.5 hours "off" time during the day.
* Patients must be able to maintain an accurate and complete diary (18-hour), with the help of a caregiver, recording "on" time, "on" time with minor dyskinesia, "on" time with troublesome dyskinesia, "off" time, and time asleep.
* Patients must be able to understand and willing to sign an approved Informed Consent form.

Exclusion Criteria:

* The patient has any indication of forms of parkinsonism other than idiopathic Parkinson's disease.
* If female, the patient is of childbearing potential, pregnant or lactating.
* The patient is in a late stage of Parkinson's disease, and is experiencing severe, disabling peak-dose or biphasic dyskinesia and/or unpredictable or widely swinging fluctuations in their symptoms.
* The patient has a current diagnosis of substance abuse (DSM-IV) or history of alcohol or drug abuse in the past 3 months.
* The patient has a current clinically significant gastrointestinal, renal, hepatic, endocrine, pulmonary or cardiovascular disease, including acute gastric ulcer, hypertension that is not well-controlled, asthma, chronic obstructive pulmonary disease (COPD), and Type I diabetes. Patients with a history of gastric ulcer who have not had an episode of acute gastritis in the last 6 months and are not currently experiencing gastric pain will be eligible for inclusion.
* The patient has second- or third-degree atrio-ventricular block or sick sinus syndrome, uncontrolled atrial fibrillation, severe or unstable angina, congestive heart failure, myocardial infarction within 3 months of the screening visit, or a significant ECG abnormality, including QTc ≥ 450 msec (males) or ≥ 470 msec (females), where QTc is based on Bazett's correction method.
* The patient has participated in a previous clinical trial with safinamide.
* The patient has a concomitant disease likely to interfere with the study medication (e.g. capable of altering absorption, metabolism or elimination of the study drug).
* The patient has a history of psychosis (e.g. schizophrenia or psychotic depression), either previously or currently, or a score ≥ 3 on Item 2 (thought disorder) or 3 (depression) of the UPDRS Section I.
* The patient has evidence of dementia or cognitive dysfunction, as indicated by a MMSE score < 22, or a score ≥ 3 on item 1 (mentation) of the UPDRS, Section I.
* The patient is depressed, as indicated by a GRID-HAMD (17-item scale) score > 17.
* The patient has a history of allergic response to anticonvulsants, levodopa, or other anti-parkinsonian agents.
* The patient has a mental or physical condition (e.g., neurotic behaviour, crippling degenerative arthritis, or limb amputation), which would preclude performing efficacy or safety assessments.
* The patient has hypersenstivity or contraindications to MAO B inhibitors.
* The patient has a current history of severe dizziness or fainting on standing, due to postural hypotension.
* The patient has a neoplastic disorder, which is either currently active or has been in remission for less than one year.
* The patient has had stereotactic surgery as a treatment for his/her Parkinson's disease.
* The patient has participated in a previous clinical trial within 30 days of entry into the study (screening visit) or has received treatment with any investigational compound within 30 days or 5 half-lives, whichever is longer, prior to screening. The use of an investigational drug other than safinamide during the study is not permitted.
* The patient is receiving treatment of his/her depression with a MAO inhibitor (e.g., selegiline), a tricyclic, or an SNRI (e.g., venlafaxine, duloxetine) at the screening visit. Note: Use of SSRIs will be permitted, provided the dose is kept as low as possible and remains stable throughout the trial.
* The patient is receiving treatment of his/her parkinsonian symptoms with a MAO inhibitor. Note: Patients receiving amantadine, COMT inhibitors, DA agonists and/or anticholinergics will be eligible to enter the trial, provided they are on a stable dose at screening.
* The patient has received treatment with any agent known to significantly inhibit or induce drug-metabolizing enyzmes (e.g., barbiturates, phenothiazines, etc.) within 4 weeks preceding the screening visit.
* The patient has received treatment with opioids (e.g., tramadol, meperidine derivatives), in the 4 weeks prior to the screening visit.
* The patient has received treatment with a depot neuroleptic within one injection cycle, or oral neuroleptics within 4 weeks prior to the screening visit. Patients who are receiving a low dose of an oral neuroleptic for treatment of psychotic symptoms (e.g., hallucinations) related to their Parkinson's disease or anti-parkinsonian medication, and who meet all other entry criteria, will be considered for enrollment, with approval of the CRO Medical Monitor. The Investigator must agree not to increase the dose of the oral neuroleptic during the trial, unless required for significant worsening.
* The patient has received treatment with a drug that has hepatotoxic potential, e.g., tamoxifen, within 4 weeks, or received radiation therapy or a drug with cytotoxic potential, e.g, chemotherapy, within one year prior to the screening visit.
* The patient has a history or a current diagnosis of HIV, tests positive for Hepatitis B surface antigen, tests positive for Hepatitis B core antibody, but negative for Hepatitis B surface antibody, or tests positive for Hepatitis C antibodies.
* The patient has any abnormality that the investigator deems to be clinically relevant, either on medical history, physical examination, ECG or a diagnostic laboratory test.
* In the judgment of the Clinical Investigator the patient is likely to be non-compliant or uncooperative during the study.
* Ophthalmologic history including any of the following conditions: albino patients, family history of hereditary retinal disease, progressive and/or severe diminution of visual acuity (i.e., 20/70), retinitis pigmentosa, retinal pigmentation due to any cause, any active retinopathy or ocular inflammation (uveitis), or progressive, severe diabetic retinopathy.

Ages: 30 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 669 (Actual)
Dates: Start 2007-01; Primary Completion 2008-10 (Actual); Study Completion 2009-02 (Actual)

PRIMARY OUTCOMES:
Increase in mean daily "on" time | baseline to endpoint
  Increase in mean daily "on" time ("on" time without dyskinesia plus "on" time with minor dyskinesia) during 18-hr diary recording period

SECONDARY OUTCOMES:
Decrease in total daily "off" time | baseline to endpoint
  Decrease in total daily "off" time, UPDRS Section III during "on" phase (based on diary) - mean change from baseline to endpoint, CGI - Change from baseline - mean score in the course of the study, change in cognition (cognitive test battery), decrease in mean "off" time following first morning dose of levodopa, improvement in the Dyskinesias Rating Scale during "on" phase, UPDRS Section II during "on" phase (based on diary),CGI- Severity of illness - mean change from baseline to endpoint, mean percent change in levodopa dose

CONTACTS AND LOCATIONS:
Overall Officials: Mohit Bhatt, MD, Principal Investigator — Jaslok Hospital, Mumbai; Neeta Mehta, MD, Principal Investigator — J.J Hospital, Mumbai; Sankhla Charulata, MD, Principal Investigator — P.D. Hinduja Hospital, Mumbai; Ajit Sowani, MD, Principal Investigator — Neurology Centre, Ahmedabad; Prosenjit Chakraborty, MD, Principal Investigator — Roby General Hospital, Kolkata; Sudhir Kothari, MD, Principal Investigator — Poona Hospital, Pune; Sunil Bandishti, MD, Principal Investigator — Ruby Hall Clinic, Pune; CU Velmurugendran, MD, Principal Investigator — Sri Ramachandra Medical College, Chennai; Suresh Kumar, MD, Principal Investigator — Vijaya Health Centre, Chennai; Devanathan Vasudevan, MD, Principal Investigator — Kamakshi Memorial Hospital, Chennai; Rupam Borgohain, MD, Principal Investigator — Nizams Institute of Medical Sciences, Hyderabad; J.K Murthy, MD, Principal Investigator — CARE Hospital, Hyderabad; Vavilikolanu Prasad, MD, Principal Investigator — Owasis Hospital & Research Centre, Hyderabad; Subashini Prabhakar, MD, Principal Investigator — Spectra Clinical Research Centre, Hyderabad; Keshava Belur, MD, Principal Investigator — J.S.S. Hospital Agrahara, Mysore; Pramod Pal, MD, Principal Investigator — NIMHANS, Bangalore; Ajit Kumar Roy, MD, Principal Investigator — St. Johns Medical College and Hospital, Bangalore; Rangashetti Srinivasa, MD, Principal Investigator — M.S. Ramaiah Memoria Hospital, Bangalore; Arun B Shah, MD, Principal Investigator — T.N.M.C and B.Y.L Nair Hospital, Mumbai; Krishnan Vijayan, MD, Principal Investigator — Kovai Medical Centre and Hospital, Coimbatore; Neeta Mehta, MD, Principal Investigator — Neeta Mehta's Clinic, Mumbai; Chandrashekhar Meshram, MD, Principal Investigator — Brain and Mind Institute, Nagpur; Nellikunja Shankar, MD, Principal Investigator — Mallikatta Neuro and Research Centre, Mangalore; Asha Kishore, MD, Principal Investigator — Sree Chitra Tirual Institute for Sciences and Technology, Kerela; Ummer Karadan, MD, Principal Investigator — Baby Memorial Hospital, Calicut; Mohammad I Sahadulla, MD, Principal Investigator — Kerala Institute of Medical Sciences, Trivandrum; Madhuri Behari, MD, Principal Investigator — All India Institute of Medical Sciences; Prahlad K Sethi, MD, Principal Investigator — Sir Ganga Ram Hospital, New Delhi; Shamsher Dwivedee, MD, Principal Investigator — Vidyasagar Institute of Mental Health and Neurosciences, New Delhi; Mukul Varma, MD, Principal Investigator — Indraprastha Apollo Hospital, New Delhi; Rajinder Bansal, MD, Principal Investigator — Dayanand Medical College and Hospital, Ludhiana; Sudesh Prabhakar, MD, Principal Investigator — Post Grad Institute of Medical Education,& Research Dept of Neurology, Chandigarh; Sunil Pradhan, MD, Principal Investigator — Institute of Human Behaviour and Allied Sciences, Dilshad Garden Delhi; Rakesh Shukla, MD, Principal Investigator — Chhatrapati Sahuji Maharaj Medical University, Lucknow; Pahari Ghosh, MD, Principal Investigator — Sri Aurbindo Seva Kendra, Kolkata; Ovidiu Bajenaru, MD, Principal Investigator — University Hospital of Emergency Hospital, Bucuresti; Cristina Panea, MD, Principal Investigator — Elias University Hospital, Bucuresti; Ana Campeanu, MD, Principal Investigator — Fundeni Hospital, Bucuresti; Marina Ticmeanu, MD, Principal Investigator — colentina Hospital, Bucuresti; Dafin Muresanu, MD, Principal Investigator — Emergency Hospital Cluj, Cluj; Angelo Bulboaca, MD, Principal Investigator — Rehabilitation Hospital Cluj, Cluj; Jozsef Szasz, MD, Principal Investigator — Emergency Hospital Targu-Mures, Targu Mures; Cristian Dinu Popescu, MD, Principal Investigator — Rehabiliation Hospital Iasi, Iasi; Mihaela Simu, MD, Principal Investigator — Emergency Hospital Timisoara no. 1, Timisoara; Dana Chirileanu, MD, Principal Investigator — Emergency Hospital Timisoara no.1, Timisoara; Roberto Eleopra, MD, Principal Investigator — Ospedale dell'Angelo, Venezia; Rocco Quatrale, MD, Principal Investigator — Arcispedale S. Anna, Ferrara; Marco Onofri, MD, Principal Investigator — Centro dell'invecchiamento, Chieti; Tanina Pia Avarello, MD, Principal Investigator — Centro di Riferimento Regionale Malattie Extra Piramidali, Palermo; Ubaldo Bonuccelli, MD, Principal Investigator — Ospedale di Viareggio, Viareggio; Giovanni Fabbrini, MD, Principal Investigator — Dip. Scienze Neurologiche, Roma; Paolo Stanzione, MD, Principal Investigator — University of Rome Tor Vergata; Fabrizio Stocchi, MD, Principal Investigator — IRCCS S. Raffaele Pisana, Roma

REFERENCES:
- See also: Related Info — http://www.newron.com/